CLINICAL TRIAL: NCT05452018
Title: Detection of Early Swallowing Time by Electromyogram and Sound Recording in Healthy Volunteers. Single-center, Prospective, Not-controlled, Not-randomized, Open-label Study.
Brief Title: Detection of Early Swallowing Time by Electromyogram and Sound Recording in Healthy Volunteers
Acronym: DEGLUTITION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); GIPSA-LAB (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC22.0096
Record Dates: First submitted 2022-06-29; First posted 2022-07-11 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
Keywords: Swallowing; Electromyogram; Intramuscular sensors; Muscular activity

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First intervention group (Experimental): Recordings of muscle activity during swallowing
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Intervention group — In healthy volunteers, activity measurement of muscles of interest by intramuscular electromyography during predefined swallowing tasks

SUMMARY:
The objective of this study is to show the feasibility of detecting the specific activity of 2 muscles during swallowing using invasive sensors in healthy volunteers.

DETAILED DESCRIPTION:
Total laryngectomy, which involves removing the larynx and performing a tracheostomy, is the standard method of surgical treatment for advanced laryngeal cancer.

It changes the patient's life and has an significant impact on his overall quality of life.

Over the last 10 years, numerous trials of artificial larynx implantation have been tested, but currently there is no method of implanting a system that detects the onset of a swallow.

The DEGLUTITION study aims to show the feasibility of detecting the specific activity of 2 muscles in swallowing using intramuscular electromyograms in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) < 25
* Affiliated with the social security plan or beneficiary of such a system
* Having signed the informed consent

Exclusion Criteria: subjects

* With chewing and/or swallowing disorders, or a history of chewing and/or swallowing disorders.
* With bleeding disorders (including patients on anticoagulants)
* With neurological disorders
* With a history of cervical surgery
* With immune deficiency
* Participating in an interventional study that may interfere with this study
* Protected person concerned by the articles L1121-5 to L1121-8 of the Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Intramuscular electromyography measurement of the activity of muscles of interest during the performance of a set of swallowing tasks. | 2 hours
  Absence or presence of visible activity on recorded signal during a swallow with the possibility to extract the TM moment (activation timing of the muscles of interest) of each muscle of interest

SECONDARY OUTCOMES:
Measurement of the TM time variable | 2 hours
  The TM time variable is assessed in milliseconds by intramuscular electromyography measurement and corresponding to activation timing of the muscles of interest
Measurement of the TS time variable | 2 hours
  Measure of TS time variable in milliseconds corresponding to passage of the food bolus through the upper esophageal sphincter. TS is assessed by signals acquired from the microphone.
Measurement of the TD time variable | 2 hours
  Measure of TD time variable in milliseconds corresponding to start of swallowing by activation of the submandibular area.TD is assessed by signals acquired from the microphone.

OTHER OUTCOMES:
Measurement of amplitude of signals for each type of swallowing and non-swallowing tasks | 2 hours
  Measure of amplitude of signals for each type of swallowing tasks (of different types of food bowls) and non-swallowing tasks (turning the head, opening the mouth, talking, smiling)
Measurement of integral of signals for each type of swallowing and non-swallowing tasks | 2 hours
  Measure of integral of signals for each type of swallowing tasks (of different types of food bowls) and non-swallowing tasks (turning the head, opening the mouth, talking, smiling)
Measurement of Root Mean Square of signals for each type of swallowing and non-swallowing tasks | 2 hours
  Measure of Root Mean Square of signals for each type of swallowing tasks (of different types of food bowls) and non-swallowing tasks (turning the head, opening the mouth, talking, smiling)

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Atallah, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Ihab Atallah, Grenoble, France

IPD SHARING:
Plan to Share IPD: No